CLINICAL TRIAL: NCT04655404
Title: A Pilot and Surgical Study of Larotrectinib for Treatment of Children With Newly-Diagnosed High-Grade Glioma With NTRK Fusion
Brief Title: A Pilot Study of Larotrectinib for Newly-Diagnosed High-Grade Glioma With NTRK Fusion
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT1903
Record Dates: First submitted 2020-11-09; First posted 2020-12-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-02

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: NTRK gene fusion; BABYPOG; HIT-SKK; Larotrectinib
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — larotrectinib

STUDY DESIGN:
Intervention Model Description: Feasibility and surgical cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Feasibility Cohort (Experimental): Larotrectinib administered PO, BID @100 mg/m2 on a 28-day cycle schedule.
  Interventions: Drug: Larotrectinib
- Surgical Cohort (Experimental): Larotrectinib administered PO, BID @100 mg/m2 3-5 days prior to definitive surgery, followed by Larotrectinib administered PO, BID @100 mg/m2 on a 28-day cycle schedule.
  Interventions: Drug: Larotrectinib; Procedure: Larotrectinib surgical

INTERVENTIONS:
Drug: Larotrectinib — 1. Larotrectinib monotherapy x2 cycles followed by disease evaluation
  2. Larotrectinib with or without chemotherapy backbone
Procedure: Larotrectinib surgical — 1. Surgical cohort: Larotrectinib x 3-5 days prior to definitive surgery followed by Larotrectinib monotherapy x2 cycles followed by disease evaluation
  2. Larotrectinib with or without chemotherapy backbone
  Arms: Surgical Cohort

SUMMARY:
This is a pilot study that will evaluate disease status in children that have been newly diagnosed high-grade glioma with TRK fusion. The evaluation will occur after 2 cycles of the medication (Larotrectinib) have been given.

The study will also evaluate the safety of larotrectinib when given with chemotherapy in your children; as well as the safety larotrectinib when given post-focal radiation therapy.

DETAILED DESCRIPTION:
In this pilot study, we will assess the disease control rate (Continued Complete Response-CCR, Complete Response-CR, Partial Response-PR and Stable Disease-SD) as well as survival rate (overall survival- OS and progression free survival- PFS) in children with newly diagnosed HGG with TRK fusion who receive 2 cycles of larotrectinib monotherapy administered orally, twice daily, at 100 mg/m2 continuously on a 28-day cycle schedule. After 2 monotherapy cycles of larotrectinib, patients with CCR or CR will continue to receive larotrectinib maintenance therapy as monotherapy for a total of 12 cycles. Continuation of treatment beyond 12 cycles, and up to 24 cycles, may be considered for patients on Larotrectinib monotherapy if they are receiving clinical benefit from the study, at the discretion of the treating physician.

Patients ≤ 48 months with PR or SD after 2 cycles of larotrectinib will go on to receive combination therapy with standard backbone chemotherapy (BABYPOG or HIT-SKK). Patients > 48 months of age (or patients ≥ 36 months of age, or patients with DIPG >18 months of age, at the discretion of the local investigator) will receive focal radiation therapy. A surgical cohort study will be explored whereby patients who have had a tumor biopsy/partial resection at their local institution and are planned to subsequently undergo definitive resection will receive 3-5 days (6-10 doses) of larotrectinib pre-surgery.

The study design of this trial requires 15 patients evaluable for disease control and for safety/ toxicity of larotrectinib as monotherapy. The surgical cohort will enroll up to 4 patients and will count towards the total 15 evaluable patients. A minimum of 6 patients will be evaluable for safety toxicity of larotrectinib in combination with standard-of-care chemotherapy or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients ≤ 21 years of age (birth to 21 years of age) at the time of study enrollment will be eligible.
* Diagnosis: Patients with newly-diagnosed high-grade (HGG), including diffuse intrinsic pontine gliomas (DIPG), whose tumors are documented in a CLIA/CAP certified lab (or clinically equivalent method considered standard in non-US sites) to harbor an NTRK fusion alteration by FISH, PCR, or next generation sequencing are eligible. Patients must have had histologically verified high-grade glioma such as anaplastic astrocytoma, glioblastoma, or H3 K27-mutant diffuse midline glioma verified at a CONNECT site.

For sites that do not have CLIA-certified equivalent (certified laboratory) to assess NTRK fusion, testing will be conducted centrally at NCH. NTRK testing will be performed by NGS using targeted RNA-sequencing (Archer Solid Tumor analysis) Please submit 10 unstained sections on charged slides at 10uM thickness, or 10 scrolls cut at 10uM thickness, along with submission of an H&E slide. Formalin-fixed paraffin embedded (FFPE) tissue block and FFPE tissue scroll specimens must contain minimum of 25% tumor Snap-frozen tissue specimens are also acceptable and they must contain a minimum of 10% tumor. Please note that turn-around time for this test is up to 21 days.

* Disease Status: Patients with disseminated DIPG or HGG are eligible only if the patient is to receive chemotherapy only, i.e. no craniospinal RT is intended to be given. MRI of spine must be performed if disseminated disease is suspected clinically by the treating physicians. Patients with primary spinal tumors are eligible only if the patient is to receive either chemotherapy or focal radiation therapy, i.e. no craniospinal RT is intended to be given. Patients with leptomeningeal disease only, with no definitive identifiable primary tumor, and documented NTRK fusion, must be discussed with the Study Chair on a case-by-case basis.
* Surgical Cohort ONLY: Patients with newly-diagnosed HGG with NTRK fusions who have undergone prior biopsy and for whom further resection is indicated for a more definitive surgery at an enrolling site will be eligible to enroll onto the surgical study. DIPG patients are not eligible for the surgical cohort.
* Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy: Patients must not have received any prior anti-cancer chemotherapy. Prior use of corticosteroids are allowed (see below Exclusion Criteria)
* Organ Function Requirements: Adequate Bone Marrow Function Defined as:

Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3 Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) Hemoglobin >8 g/dL (may receive transfusions)

- Adequate Renal Function Defined as: Serum creatinine within normal institutional limits, or Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2

- Adequate Liver Function Defined as: Total bilirubin ≤ 2.5 × institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional upper limit of normal

- Adequate Pulmonary Function Defined as: Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest).

- Adequate Neurologic Function Defined as: Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled. See Section 5.5.2 and Appendix III for EIAED guidelines.

- Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Concomitant Medications Investigational Drugs: Patients who have previously received or are currently receiving another investigational drug are not eligible.

Anti-cancer Agents: Patients who have previously received or are currently receiving other anti-cancer agents, including chemotherapy, immunotherapy, monoclonal antibodies, biologic or targeted therapy, are not eligible

* Infection: Patients must not have any active, uncontrolled systemic bacterial, viral or fungal infection.
* Patients who have received prior solid organ transplantation are not eligible.
* Patients must not have malabsorption syndrome or other condition affecting oral absorption.
* Patients must not be receiving any treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducer. (See Appendix III.) Strong inducers or inhibitors of CYP3A4 should be avoided from 7 days prior to enrollment to the end of the study.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | At the end of Cycle 2 (each cycle is 28 days)
  To assess the disease control rate (Complete Response [CR], Continued Complete Response [CCR], Partial Response [PR] and Stable Disease [SD]) of larotrectinib in young children newly diagnosed with HGG carrying NTRK fusion after 2 cycles of larotrectinib monotherapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From Day 1 of treatment through 30 days following end of protocol treatment
  To assess the safety and tolerability of larotrectinib given in combination with chemotherapy or post-focal radiation therapy in young children newly diagnosed with HGG carrying NTRK fusion. This will be achieved by calculating the number of participants with, as well as frequency and severity of, larotrectinib-related Adverse Events as assessed by CTCAE v5.0.
Maximum Plasma Concentration [Cmax] of larotrectinib | Days 1 through 5 of surgical cycle
  To characterize the plasma pharmacokinetics (PK) of larotrectinib in children newly diagnosed with HGG carrying NTRK fusions who undergo a second definitive resection. This will be achieved by measuring the Maximum Plasma Concentration (Cmax) of larotrectinib in blood (plasma) samples collected at pre-dose (day -5), pre-surgery (day -1) and during surgery.
Tumor Concentration of larotrectinib | Day 5 of surgical surgical cycle
  To characterize the tumor pharmacokinetics (PK) of larotrectinib in children newly diagnosed with HGG carrying NTRK fusions who undergo a second definitive resection by measuring the concentration of larotrectinib in tumor tissue collected on day 5 of surgical cycle

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  To assess the objective response rate (ORR) (Complete Response [CR] and Partial Response [PR]) of larotrectinib in children newly-diagnosed with HGG carrying NTRK fusion after 2 cycles of larotrectinib monotherapy.
Survival rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To assess overall (OS) and progression-free survivals (PFS) of children newly diagnosed with HGG carrying NTRK fusion treated with a larotrectinib-containing regimen at 1, 3 and 5 years and compared to historical data from BABYPOG and HIT-SKK.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chi, MD, Study Chair — Dana Farber/ Boston Children's Cancer and Blood Disorders Center; Maryam Fouladi, MD, Study Chair — Nationwide Children's Hospital
Locations (21):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Germany (5):
  - Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg
  - University Medical Center Augsburg, Augsburg
  - University Hospital Berlin, Berlin
  - University Hospital Koln, Cologne
  - University Medical Center Gottingen, Göttingen
- Starship Children's Hospital, Auckland, Grafton, New Zealand